CLINICAL TRIAL: NCT01644968
Title: Phase 1 Trial of a Monoclonal Antibody to OX40 in Patients With Advanced Cancer.
Brief Title: Phase 1 Study of Anti-OX40 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-066A
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Advanced Cancer
Keywords: metastatic carcinoma; lymphoma; sarcoma; anti-OX40
MeSH Terms: conditions — Carcinoma; Lymphoma; Sarcoma | interventions — Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KLH + anti-OX40 (Experimental): Day 1: KLH + anti-OX40; Day 3: anti-OX40; Day 4: anti-OX40; Day 29: Tetanus vaccine
  Interventions: Drug: Cohort 1 anti-OX40; Drug: Cohort 2 anti-OX40; Drug: Cohort 3 anti-OX40; Biological: Tetanus Day 29; Biological: KLH Day 1
- Tetanus vaccine + anti-OX40 (Experimental): Day 1: Tetanus vaccine + anti-OX40; Day 3: anti-OX40; Day 5: anti-OX40; Day 29: KLH
  Interventions: Drug: Cohort 1 anti-OX40; Drug: Cohort 2 anti-OX40; Drug: Cohort 3 anti-OX40; Biological: Tetanus Day 1; Biological: KLH Day 29

INTERVENTIONS:
Drug: Cohort 1 anti-OX40 — 0.1 mg/kg anti-OX40 on days 1, 3, and 5
Drug: Cohort 2 anti-OX40 — .4 mg/kg anti-OX40 on days 1, 3, and 5
Drug: Cohort 3 anti-OX40 — 2.0 mg/kg anti-OX40 on days 1, 3, and 5
Biological: Tetanus Day 29 — Tetanus toxoid vaccine 0.5ml (5 LF/ml tetanus toxoid)on Day 29
  Other Names: Tetanus Toxoid, Tetanus Toxoid Adsorbed
  Arms: KLH + anti-OX40
Biological: Tetanus Day 1 — Tetanus toxoid vaccine 0.5ml (5 LF/ml tetanus toxoid)on Day 1.
  Other Names: Tetansu Toxoid, Tetanus Toxoid Adsorbed.
  Arms: Tetanus vaccine + anti-OX40
Biological: KLH Day 1 — 1 mg KLH in 1 cc diluent subcutaneously on Day 1.
  Other Names: Immucothel.
  Arms: KLH + anti-OX40
Biological: KLH Day 29 — 1 mg KLC in 1 cc diluent by subcutaneous injection on Day 29.
  Other Names: Immucothel.
  Arms: Tetanus vaccine + anti-OX40

SUMMARY:
This study is designed to determine the safety and highest tolerated dose of anti-OX40 in patients with advanced cancer.

DETAILED DESCRIPTION:
This study will evaluate the safety and determine the maximal tolerated dose of anti-OX40; evaluated the immune response to the study treatment; measure the pharmacokinetics of anti-OX40; monitor tumor regression, and identify the most biologically active dose of anti-OX40 to induce antigen-specific responses to a variety of immunogens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncurable metastatic carcinoma, lymphoma, or sarcoma.
* ECOG performance status 0, 1, 2
* No active bleeding
* No clinical coagulopathy
* Anticipated lifespan greater than 12 weeks

Exclusion Criteria:

* Active residual toxicity from prior therapies
* Active Infection
* HIV positive
* Hepatitis B or C positive
* Pregnant or nursing women
* Requirement for oral steroids
* Brain metastases
* Presence or history of autoimmune disease
* Shellfish or tetanus allergy
* Splenomegaly
* Lymph nodes greater than 10 cm in maximal diameter
* Uncontrolled angina or class II or IV heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-11 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 28 Days
  A dose limiting toxicity is defined as any grade >=3 hematologic (except lymphopenia) or non-hematologic toxicity (except hypothyroidism or vitiligo) that, in the opinion of the investigator is considered at lease possibly related to the study treatment. If DLT is observed in greater than two patient in any cohort, then the previous cohort will be the maximal tolerated dose.

SECONDARY OUTCOMES:
Immune Response | Pre-study, Days 5, 8, 15, 29, 36, 43, and 57.
  Blood tests and leukapheresis product will be collected to determine the response to three types of reporter antigens: (1) new antigen (keyhole limpet hemocyanin (KLH)), (2) recall protein antigen (tetanus), and (3) viral antigen (cytomegalovirus (CMV)). Changes in the number of antigens will be used to determine immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Cancer Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curti BD, Kovacsovics-Bankowski M, Morris N, Walker E, Chisholm L, Floyd K, Walker J, Gonzalez I, Meeuwsen T, Fox BA, Moudgil T, Miller W, Haley D, Coffey T, Fisher B, Delanty-Miller L, Rymarchyk N, Kelly T, Crocenzi T, Bernstein E, Sanborn R, Urba WJ, Weinberg AD. OX40 is a potent immune-stimulating target in late-stage cancer patients. Cancer Res. 2013 Dec 15;73(24):7189-7198. doi: 10.1158/0008-5472.CAN-12-4174. Epub 2013 Oct 31. PMID 24177180